CLINICAL TRIAL: NCT02036398
Title: Comparison of Complications Between Patients Undergoing Standard Percutaneous Nephrolithotomy With Nephrostomy Tube Placement and Tubeless Percutaneous Nephrolithotomy With Double J Stent Only Placement
Brief Title: Tubeless Versus Standard Upper Pole Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Hanan Goldberg, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RMC-6405
Record Dates: First submitted 2014-01-10; First posted 2014-01-15 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Pleural Effusion
Keywords: Percutaneous Nephrolithotomy (PCNL); Nephrostomy; Double J stent; PleuraL Effusion
MeSH Terms: conditions — Pleural Effusion | interventions — Nephrotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nephrostomy tube + double J stent (Active Comparator): Standard therapy group with nephrostomy tube and double J stent left at the end of the PCNL
  Interventions: Device: Double J stent without nephrostomy; Device: nephrostomy tube and double J stent
- Double J stent without nephrostomy (Experimental): Double J stent only left at the end of the procedure
  Interventions: Device: Double J stent without nephrostomy

INTERVENTIONS:
Device: Double J stent without nephrostomy — Double J stent only left at the end of the procedure without placement of a nephrostomy tube
Device: nephrostomy tube and double J stent — Double J stent and nephrostomy tube left at end of procedure
  Arms: Nephrostomy tube + double J stent

SUMMARY:
Comparison of complications between standard upper pole percutaneous nephrolithotomy (PCNL) with nephrostomy placement and double J stent and PCNL with double J placement only without nephrostomy.

DETAILED DESCRIPTION:
Measurement of complications in and comparison between two groups of patients undergoing upper pole PCNL. First group consists of patients left with nephrostomy and double J stent and the second group includes patients left with double J stent only without nephrostomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing upper pole percutaneous nephrolithotomy older than 18 years of age and willing to participate

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients unwilling to participate in the study
* Patients that nephrostomy tube placement was a prerequisite at the end of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with pleural effusion | 30 days
  Assessment and comparison of pleural effusion incidence between patients in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Goldberg, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Urology department, Rabin Medical Center, Petach Tiqva, Israel

REFERENCES:
- [Derived] Goldberg H, Nevo A, Shtabholtz Y, Lubin M, Baniel J, Margel D, Ehrlich Y, Lifshitz D. Tubeless supra-costal percutaneous nephrolithotomy is associated with significantly less hydrothorax: a prospective randomized clinical study. BJU Int. 2020 Feb;125(2):276-283. doi: 10.1111/bju.14950. Epub 2019 Dec 3. PMID 31721407